CLINICAL TRIAL: NCT05666752
Title: A 8 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Allium Cepa L. Peel Heated Water Extract on Immunity Enhancement
Brief Title: Effect of Intake of Allium Cepa L. Peel Heated Water Extract on Immunity Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yongsoon Park, Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NAS-IE-ON
Record Dates: First submitted 2022-12-13; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Upper Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allium Cepa L. Peel Heated Water Extract (Experimental): 4 capsules/day after meal(1,200 mg/day) for 8 weeks
  Interventions: Dietary Supplement: Allium Cepa L. Peel Heated Water Extract
- Placebo (Placebo Comparator): 4 capsules/day after meal(1,200 mg/day) for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Allium Cepa L. Peel Heated Water Extract — 4 capsules/day after meal(1,200 mg/day) for 8 weeks
  Arms: Allium Cepa L. Peel Heated Water Extract
Dietary Supplement: Placebo — 4 capsules/day after meal(1,200 mg/day) for 8 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Allium Cepa L. Peel Heated Water Extract on Immunity Enhancement

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled human trial. 40 subjects were randomly divided into Allium Cepa L. Peel Heated Water Extract or a placebo group. Immunity Enhancement profiles before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-75 years
* Symptoms of upper respiratory infection at least once within past 12 months

Exclusion Criteria:

* Cardio-cerebrovascular, endocrine, immune, respiratory, musculoskeletal, inflammatory, hematologic, tumorigenic, gastrointestinal diseases, etc.
* Vaccination within past 2 months
* BMI < 18.5 kg/m2 or 35 kg/m2 ≤ BMI
* Immunity enhancement agents within past one months
* Allergic or hypersensitive to any of the ingredients in the test products
* Antipsychotic drugs therapy within past 3 months
* History of alcoholism or drug abuse
* Participation in any other clinical trials within past 3 months
* Pregnant or lactating women
* Judged ineligible to participate in the trial by the principal investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Changes of Natural killer(NK) cell activity | At week 0 and week 8
  Changes of Natural killer(NK) cell activity will be assessed before and after the intervention.
  PBMCs were isolated by density gradient separation, resuspended in phosphate-buffered saline, and determined using trypan blue solution. Natural killer(NK) cell activity was calculated from the results of nonradioactive cytotoxicity assay kits. Effector cells (PBMCs) were seeded in 96-well plates, with 50 ul of target cells (K562), incubated for 4 hours. cytotoxicity was calculated using the following formula: [(experimental-effector spontaneous-target spontaneous)/(target maximum-target spontaneous)]*100.

SECONDARY OUTCOMES:
Changes of Cytokines(INF-gamma, Interleukin(IL)-2, IL-6, IL-12, Tumor Necrosis Factor(TNF)-alpha, and IL-1beta) | At week 0 and week 8
  Changes of Cytokines(INF-gamma, IL-2, IL-6, IL-12, TNF-alpha, and IL-1beta) will be assessed before and after the intervention.
  the serum levels of cytokines, including INF-gamma, IL-2, IL-6, IL-12, TNF-alpha, and IL-1beta will be measured.
Changes of Wisconsin Upper Respiratory Symptom Survey-21 | At week 0 and week 4 and week 8
  Changes of Wisconsin Upper Respiratory Symptom Survey-21 will be assessed before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yongsoon Park, Ph.D., Principal Investigator — Hanyang University
Locations (1):
- Hanyang University, Seoul, South Korea

REFERENCES:
- [Derived] Cho H, Kim S, Lee SH, Park Y. Effect of onion (Allium cepa L.) peel extract on natural killer cell and cytokines in a randomized, double-blind, placebo-controlled trial. Nutr Res Pract. 2024 Feb;18(1):33-45. doi: 10.4162/nrp.2024.18.1.33. Epub 2024 Jan 11. PMID 38352207